CLINICAL TRIAL: NCT04877834
Title: A Single Center, Open Label, Randomized, Single-dose, Two-period, Two-way Cross-over Study to Compare the Rate and Extent of Absorption of DelanzoᵀᴹDR 60mg (Dexlansoprazole) Capsule With Dexilant® 60mg (Dexlansoprazole) Capsule in Healthy Pakistani Subjects.
Brief Title: Bioequivalence Study of DelanzoᵀᴹDR 60mg (Dexlansoprazole) Capsule With Dexilant® 60mg (Dexlansoprazole) Capsule in Healthy Pakistani Subjects.
Acronym: BABE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: SAMI Pharmaceuticals (Pvt.) Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-035-DEX(D)-2020
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Bioequivalence Study
Keywords: Bioequivalence Study, Healthy Pakistani Population,; Dexlansoprazole Capsule
MeSH Terms: interventions — Dexlansoprazole; Capsules; Hardness

STUDY DESIGN:
Intervention Model Description: A single center, open-label, randomized, single-dose, two-period, two-way, cross-over study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DelanzoTMDR group (Experimental): Subjects will take DelanzoTMDR 60 mg Capsule, manufactured by SAMI Pharmaceuticals (Pvt.) Ltd. after at least 10 hours' fast, with 240 mL of ambient temperature water at their scheduled dosing time-point.
  Interventions: Drug: Dexlansoprazole
- Dexilant® Group (Active Comparator): Subjects will take Dexilant® 60 mg Capsule, manufactured by Takeda Pharmaceutical Company Limited after at least 10 hours' fast, with 240 mL of ambient temperature water at their scheduled dosing time-point.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole capsule prepared by SAMI Pharmaceuticals will be administered to this arm.
  Other Names: DelanzoTMDR 60 mg capsule, hard
  Arms: DelanzoTMDR group
Drug: Dexlansoprazole — Dexlansoprazole capsule prepared by Takeda Pharmaceutical Company will be administered to this arm.
  Other Names: Dexilant® 60 mg capsule, hard
  Arms: Dexilant® Group

SUMMARY:
Single oral dose of study drug in two period(s) separated by a washout period of seven (07) days. Blood samples will be taken up to 24.0 hours post-dose.

DETAILED DESCRIPTION:
Test Product DelanzoTMDR 60 mg Capsule, manufactured by SAMI Pharmaceuticals (Pvt.) Ltd.or Reference Product Dexilant® 60 mg Capsule, manufactured by Takeda Pharmaceutical Company Limited. will be administered to healthy male Pakistani volunteers with 240 mL ambient temperature water and blood samples will be taken up to 24 hours post dose for the calculation of Cmax, Tmax, AUC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 55 years inclusive.
* Subjects with a body mass index (BMI) from 18.5 to 30 kg/m2.
* Subject is able to fast for 14 hours and consume standard meals.
* Subjects who are healthy as determined by routine physical examination, including vital sign monitoring (i.e., blood pressure, heart rate, and temperature), 12-Lead ECG, and safety laboratory analysis (i.e., hematology, blood biochemistry, and urinalysis) or viral serology as determined by the investigator.
* Subjects should have negative urine test for drugs of abuse (morphine & cannabinoids will be tested) and alcohol breath analysis at screening and prior to each check-in.
* Subjects who are able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study check-In day.
* Subject agreed not to consume food or beverages including tea, coffee, cola drinks, chocolates containing xanthine derivatives (including caffeine, theobromines, etc.) and/or poppy seeds (Khash khash) within 48 hours prior to drug administration until last blood draw in each study period.
* Subject agreed not to intake prescription drugs (especially any other PPI, Antiretroviral (e.g. rilpivirine, atazanavir and nelfinavir), Warfarin, clopidogrel, methotrexate, drugs dependent on gastric pH for absorption, etc.) within 14 days or 5 half-lives (whichever is longer) prior to first dose of study medicine.
* Subject agreed not to intake non-prescription drugs (OTC) within 14 days prior to first dose of study medicine.
* Subject agreed to discontinue vitamins, dietary and herbal supplements within 14 days prior to the first dose of study medication.
* Subject agreed not to consume grapefruit and/or its products within 14 days prior to the start of study.

Exclusion Criteria:

* Subjects who refused to sign Informed Consent Form.
* Inability to take oral medication.
* Pregnant and lactating females.
* History of smoking ≥3 cigarette/day, alcoholism, and positive test for drug of abuse, heavy pan or gutka user as judged by teeth / mouth inspection.
* Subject has clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
* Subjects allergic to Dexlansoprazole and/or other Antacid drugs.
* Subject has received any investigational drug within four weeks.
* Participated in any clinical trials within 3 months.
* Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
* History of any significant illness in the last four weeks which might confound in the result of the study or post additional risk in administrating Dexlansoprazole to the subject.
* Subjects tested positive for syphilis (VDRL) or is known to have serum hepatitis or carrier of the Hepatitis B surface antigen (HBs Ag) or are carriers of antibodies to hepatitis C virus (anti-HCV) or to the human immunodeficiency virus (HIV-1 or HIV-2).
* Subject tested positive for COVID-19 or is known to have such family members who tested positive for COVID-19 in recent times.
* Subject has undergone any major surgery within 3 months prior to the start of the study, unless deemed eligible, otherwise by the Principal Investigator or whomever he/she may designate.
* Subject has a condition, which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or elimination of drugs.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of asthma, anaphylaxis or anaphylactic reactions, severe allergic responses.
* A heart rhythm disorder (especially if you take medication to treat it) or history of long QT syndrome.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Pakistani Population
Enrollment: 60 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Cmax | 24 hours
  Determination of plasma drug concentration
Tmax | 24 hours
  Time to reach maximum plasma drug concentration
AUC | 24 hours
  Area under the Plasma concentration Versus time curve

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — Center for bio-equivalence, and clinical research, university of karachi; Dr. Naghma Hashmi (Co-PI), PhD, Principal Investigator — Center for bio-equivalence, and clinical research, university of karachi
Locations (1):
- Center for Bioequivalence Studies and clinical research, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will only be available upon reasonable request to PI, subject to the confidentiality of the participants.